CLINICAL TRIAL: NCT00735254
Title: Pulsed Dye Laser and Affirm Laser in the Treatment of Abdominoplasty Scars
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI decision
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 08-352
Record Dates: First submitted 2008-08-13; First posted 2008-08-14 (Estimated); Results first posted 2018-02-08 (Actual); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Abdominoplasty Scars
Keywords: post; surgical
MeSH Terms: interventions — Lasers, Dye

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Pulsed dye laser (Active Comparator): PDL Patient will be have scar treated with pulsed dye laser.
  Interventions: Device: pulsed dye laser
- Affirm laser (Active Comparator): Patient will be have scar treated with Affirm Laser
  Interventions: Device: Affirm Laser
- combined PDL and Affirm Lasers (Active Comparator): Patient will be have scar treated with combined Affirm + PDL
  Interventions: Device: combined PDL and Affirm Lasers
- Placebo (Placebo Comparator): Patient will be have scar treated with Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Device: pulsed dye laser — patient will have scar treated with pulsed dye laser
  Other Names: VBEAM
  Arms: Pulsed dye laser
Device: Affirm Laser — patient will have scar treated with Affirm laser
  Other Names: non-ablative laser
  Arms: Affirm laser
Device: combined PDL and Affirm Lasers — patient will have scar treated with Affirm and pulsed dye lasers
  Other Names: VBEAM, non-ablative laser
  Arms: combined PDL and Affirm Lasers
Other: Placebo — patient will receive no treatment
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the effect of using a pulsed dye laser (the VBEAM), a non-ablative laser (the Affirm) and a combination of both lasers to improve the appearance of your surgical scar. Both the pulsed dye laser and Affirm laser are approved by the US Food and Drug Administration (FDA) for the treatment of scars. Surgical scars are a type of scar that can benefit from laser therapy. Redness and the appearance of small blood vessels near the surface of the skin (telangiectasias) develop in such scars as part of the normal healing process and usually spontaneously remit, but often slowly and incompletely. In many cases, lasers can accelerate the clearing of this redness and also improve scar texture.

DETAILED DESCRIPTION:
In summary, we will perform a total of three laser treatments. A personal interview, clinical examination, and a photograph will be taken at each visit. At the end of the three treatments, a final personal interview, clinical evaluation and photograph will be taken to document the effects of the laser treatments. At the end of the study, the patient will have the option to receive two additional laser treatments four weeks apart, also at no cost, to the entire scar.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* No significant medical illness
* Surgical procedure that involves closure of the transverse abdominal incision performed in the department of dermatology and plastic surgery at the Cleveland Clinic main campus.
* Subjects with the willingness and ability to understand and provide informed consent

Exclusion Criteria:

* Under 18 years of age
* Pregnancy or Lactation
* Subjects currently taking blood thinners or who have had chemotherapy or radiation within the last 6 months
* Subjects with liver/kidney disease, diabetes mellitus, hypertension, connective tissue disease or who are immunocompromised
* Subjects with a known susceptibility to keloid formation or hypertrophic scarring
* Subjects who are unable to understand the protocol or to give informed consent
* Subjects with mental illness
* Subjects with obvious non-healing wound

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-07; Primary Completion 2009-07 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Tung, MD, Study Director — The Cleveland Clinic
Locations (1):
- Cleveland Clinical Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pulsed Dye Laser | Affirm Laser | Combined PDL and Affirm Lasers | Placebo
Started | 1 | 1 | 1 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 1 | 0
Not completed — Protocol Violation | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: PI left institution, no data available.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pulsed Dye Laser | Affirm Laser | Combined PDL and Affirm Lasers | Placebo | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
Age, Customized — PI left institution, no data available. Population: PI left institution, no data available.
Sex/Gender, Customized — PI left institution, no data available. Population: PI left institution, no data available.

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of PDL vs Affirm Laser vs Combined Laser Treatments in Appearance of Surgical Scar
Description: The purpose of this study is to determine the efficacy of the 585-nm pulsed dye laser (PDL) and 1440-nm Affirm laser in the treatment of surgical scars starting one week after closure of transverse abdominal incision.
Time Frame: 1 year
Population: study was not conducted per protocol, data was not collected, study terminated. Reported to IRB and closed study.
Arm/Group | Pulsed Dye Laser | Affirm Laser | Combined PDL and Affirm Lasers | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: protocol was not followed and data was not collected. reported to IRB, closed study. PI left institution
Description: protocol was not followed and data was not collected. reported to IRB, closed study. PI left institution
Arm/Group | Pulsed Dye Laser | Affirm Laser | Combined PDL and Affirm Lasers | Placebo
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
protocol was not followed and data was not collected. reported to IRB, closed study. PI left institution

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes